CLINICAL TRIAL: NCT05193539
Title: Effects of Comprehensive Augmented and Virtual Reality for Upper Limb Rehabilitation in First-Ever Stroke Patients
Brief Title: Effects of Comprehensive Augmented and Virtual Reality in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Geol Do, M.D, PhD, Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-07-012-021
Record Dates: First submitted 2021-12-09; First posted 2022-01-18 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: Virtual Reality; Augmented Reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded study. Individuals were randomly assigned to either the experimental group or control group using a computer-generated randomization technique. The randomization list was created on blocks of four and generated at the start of the study using a computerized program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher responsible for randomization was independent from the assessors, assuring blindness to treatment allocation and randomization procedures. The blinded assessor performed the baseline and post-treatment assessments. The patients and the occupational therapists were not blinded due to the nature of treatment modality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented reality and virtual reality rehabilitation (Experimental): This group underwent augmented reality and virtual reality rehabilitation for 60 minutes per session, 5 days per week for 2 weeks.
  Interventions: Behavioral: Augmented reality and virtual reality rehabilitation
- Conventional occupational therapy (Active Comparator): This group underwent conventional occutational therapy for 60 minutes per session, 5 days per week for 2 weeks.
  Interventions: Behavioral: Conventional occupational therapy

INTERVENTIONS:
Behavioral: Augmented reality and virtual reality rehabilitation — This group underwent augmented reality and virtual reality rehabilitation with 4 different systems.
  The RAPAEL Smart Glove® is a wearable sensory system that contains a single 9-axis movement and position sensor with 3 acceleration channels, 3 angular rate channels, and 3 magnetic field channels that measures wrist movements, and 5 bending sensors that measure finger movements. The RAPAEL Smart Board® is a rehabilitation system used to improve arm function by practicing gravity-compensated movements. The RehabMaster® is a game-based Kinect sensor AR rehabilitation system which uses a 3D camera to digitize patient movements and quickly analyze their range of motion, speed, motion angle, and movement cycles. rehabilitation exercise using games to encourage active arm and trunk movements and promote successful rehabilitation. The COG-Trainer® is a VR system that uses a training device synchronized with the screen through simulation.
  Arms: Augmented reality and virtual reality rehabilitation
Behavioral: Conventional occupational therapy — The group underwent standard ocupational therapy, such as range of motion and strengthening exercises for the affected upper extremity, table-top activities, and training for activities of daily living.
  Arms: Conventional occupational therapy

SUMMARY:
The purpose of this study was to assess the efficacy of augmented and virtual reality-based rehabilitation programs on improving upper extremity function in subacute stroke patients.

DETAILED DESCRIPTION:
This was a randomized, single-blinded study, conducted at a single acute rehabilitation unit in a university hospital. In this study, the effect of augmented and virtual reality-based rehabilitation for the recovery of subacute stroke patients compared with conventional occupational therapy was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* First ever stroke
* Onset of stroke less than 3 months
* Sufficiently medically stable to participate in active rehabilitation
* Mild-to-moderate upper extremity motor impairments (Brunnstrom stage for the upper extremity 2-6).

Exclusion Criteria:

* Severe cognitive impairment (defined as score < 10 on the Mini-Mental State Examination)
* Evidence of apraxia
* Clinical history of neglect
* Previous upper extremity hemiplegia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity score | Baseline
  range (0-126), higher scores mean a better motor function
Fugl-Meyer Assessment for Upper Extremity score | 2 weeks after intervention
  range (0-126), higher scores mean a better motor function

SECONDARY OUTCOMES:
Box and Block Test | Baseline
  higher scores mean a worse motor function
Box and Block Test | 2 weeks after intervention
  higher scores mean a worse motor function
Modified Barthel Index | Baseline
  range (0-100), higher scores mean a better activity of daily living
Modified Barthel Index | 2 weeks after intervention
  range (0-100), higher scores mean a better activity of daily living
Motor Activity Log of Amount of Use and Quality of Movement | Baseline
  range (0-150), higher scores mean a better activity of daily living
Motor Activity Log of Amount of Use and Quality of Movement | 2 weeks after intervention
  range (0-150), higher scores mean a better activity of daily living
EuroQol Visual Analogue Scale | Baseline
  range (0-100), higher scores mean a better quality of life
EuroQol Visual Analogue Scale | 2 weeks after intervention
  range (0-100), higher scores mean a better quality of life
Berg Balance Scale | Baseline
  range (0-56), higher scores mean a better balance function
Berg Balance Scale | 2 weeks after intervention
  range (0-56), higher scores mean a better balance function
Grip strength (kg) | Baseline
  higher scores mean a better hand function
Grip strength (kg) | 2 weeks after intervention
  higher scores mean a better hand function
Hand response reaction time | Baseline
  higher scores mean a worse hand function
Hand response reaction time | 2 weeks after intervention
  higher scores mean a worse hand function

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea